CLINICAL TRIAL: NCT03881384
Title: Early Evaluation of Circulating Tumor DNA as Marker of Therapeutic Efficacy in Breast Cancer Patients During Neoadjuvant Chemotherapy
Brief Title: Circulating Tumor DNA as Marker of Therapeutic Efficacy in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2018-001
Record Dates: First submitted 2019-03-17; First posted 2019-03-19 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Breast Neoplasms
Keywords: ctDNA
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor biopsy specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ctDNA level: ctDNA level during neoadjuant chemotherapy
  Interventions: Other: ctDNA level during neoadjuant chemotherapy

INTERVENTIONS:
Other: ctDNA level during neoadjuant chemotherapy — Draw blood from each enrolled patient every time before chemotherapy and measure the ctDNA level in plasma.

SUMMARY:
In nonmetastatic local advanced breast cancer patients, we are going to investigate whether circulating tumor DNA (ctDNA) detection can reflect the tumor response to neoadjuvant chemotherapy (NCT) and detect minimal residual disease after surgery.

DETAILED DESCRIPTION:
Breast cancer is the most common malignant tumor in women worldwide, and chemotherapy is still the main method of breast cancer treatment. And for locally advanced breast cancer patients, neoadjuvant chemotherapy can further improve treatment efficacy, improve prognosis and increase the rate of breast conserving surgery. The persistence of a minimal residual disease at distant sites after the treatment of a localized breast cancer is a key parameter for posttreatment survival but cannot be reliably assessed by the current biological or radiological tools. Therefore, the prediction of the chemotherapy efficacy is very important. ctDNA, corresponds to fragmented DNA released into the blood stream by tumor masses, the detection and quantification of circulating tumor DNA (ctDNA) is a very promising tool that can assess tumor burden, response to therapy, and minimal residual disease. In this study, we wil collect breast cancer cases treated with neoadjuvant chemotherapy, draw blood and evaluate the efficacy each time before chemotherapy and after surgery, then measure the concentration of ctDNA in each sample. We will also analyze the demographic data,basic treatment and follow-up data including relapse, metastasis and survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients pre- or post-menopausal must have histologically confirmed early stage/locally advanced invasive breast cancer;
* Tumor size ≥ 0.5cm (clinical or radiographic measurements);
* Any nodal status allowed;
* Age > 18 years old;
* Felt to be a possible candidate for neoadjuvant systemic therapy by their treating physician;
* ECOG score<=2;

Exclusion Criteria:

* Known metastatic disease;
* With serious heart, lung, liver diseases;
* Poor cardiac function;
* Pregnant;
* Patients with other malignant tumor or treated before;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are considered possible candidates for neoadjuvant chemotherapy, by clinical-pathologic features.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The concentration of circulating DNA(ctDNA) | From date of neoadjuvant chemotherapy decided until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Take the blood each time before chemtherapy and measure the concentration of ctDNA

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun He, PhD, Principal Investigator — First Affiliated Hospital of Xian Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No